CLINICAL TRIAL: NCT04233554
Title: Implementation and Evaluation of Patient Priorities Care-North Carolina for Older Adults With Multiple Chronic Conditions
Brief Title: Patient Priorities Care-North Carolina
Acronym: PPC-NC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to identify enough practices and clinicians to participate in the study.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Yale University (Other); North Carolina Translational and Clinical Sciences Institute (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-2380; R01AG062686 (NIH)
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Multiple Chronic Conditions
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - Implementing Patient Priorities Care (Experimental): Practice staff and providers will be trained on how to identify patient health priorities. Staff and clinicians will implement Patient Priorities Care, document priorities in EHRs, and align patient priorities with health care decisions.
  Interventions: Behavioral: Patient Priorities Care
- Control Arm (No Intervention): Control arm practices will receive no intervention and patients will receive usual care.

INTERVENTIONS:
Behavioral: Patient Priorities Care — Patients will participate in a structured conversation in which the facilitator (i.e. social worker) helps patients identify their health goals, measurable, actionable, realistic outcomes (e.g. walk ½ mile daily). Both practice and patient level data will be collected.
  Arms: Intervention Arm - Implementing Patient Priorities Care

SUMMARY:
The long-term goal of this research is to re-engineer clinical decision-making for older adults with multiple chronic conditions (MCC) to focus on patients' self-identified health priorities. The overall objective of this study is to implement and evaluate an intervention called Patient Priorities Care (PPC) intervention with 20 primary care clinicians in North Carolina (NC), using a hybrid effectiveness-implementation design. Guided by the Minimally Disruptive Medicine model, the central hypothesis is that clinical decision-making guided by patients' priorities will result in less burdensome care for patients and their families, increase patient goal setting, facilitate patient-provider shared decision-making, and improve patient quality of life and satisfaction with care. As the prevalence, costs, and treatment burden of MCC continue to rise, new approaches to care are urgently needed in this growing population. Findings from this study will inform practical approaches for aligning clinical decision-making in older adults with MCC with their health priorities.

DETAILED DESCRIPTION:
Multiple chronic conditions (MCC) among older adults are prevalent and costly. Almost 70% of Americans 65 years and older, most of whom are Medicare beneficiaries, have at least two chronic medical conditions and 14% have 6 or more chronic conditions, which lowers life expectancy and reduces quality of life (QOL). Over 90% of the Medicare spending is devoted to individuals with MCC. Despite these facts, health care and research are primarily focused on single diseases. Living with MCC is complex and burdensome. Individuals with MCC are burdened by the work required to manage their illnesses. This work includes processing complex and sometimes conflicting information about symptoms and treatments, integrating clinician recommendations into their daily lives, monitoring their disease and managing symptoms and medications, enlisting support from others, and coordinating and following-through with frequent clinician visits. Family members are intimately involved in supporting health-related behaviors of individuals with MCC. On average, patients with MCC and their family caregivers spend 2 hours a day on health-related activities plus an additional 2 hours for every visit to a health care facility (between travel time, wait time, and actual time receiving the health service). Medicare patients see, on average, 2 primary care clinicians and 5 specialists annually. Attending frequent clinician visits increases treatment burden for these patients, independent of the actual treatments received. This fragmented provision of health care for older adults with MCC and their family members requires a simplified, coordinated approach to care that reduces burden on patients and families.

Patient priorities care (PPC) is an innovative solution to address the discrepancy between the care older adults with MCC receive and the outcomes they want. When faced with tradeoffs between desired QOL outcomes and health care options that can increase treatment burden, individuals vary in their health priorities. Patients' health priorities include both their health outcome goals and their health care preferences. Health outcome goals are the personal health and life outcomes that patients hope to achieve through their health care (i.e., function, survival, social activities, or symptom relief). To inform clinical decision-making, health outcome goals should be specific, measurable, actionable, realistic, and time-bound (SMART) and aligned with what matters most to patients (patients' values). The overall goal is to evaluate effectiveness and implementation of PPC- an approach to clinical decision-making that is used by patients' existing clinical care team members, in North Carolina. The feasibility and efficacy of this approach has previously been demonstrated in a large primary care practice in Connecticut.

The investigators will randomize 20 primary care clinicians to PPC-NC or usual care (UC). Clinicians randomized to UC will not receive the PPC-NC intervention.

The PPC process begins when a 'facilitator' (i.e. an individual with motivational interviewing skills) meets with the patient and helps patients identify their value-based priorities during a structured conversation. Values, which represent what matters most to individuals, tend to remain stable over time and form the basis of patients' health outcome goals. Patients' values are clarified using questions such as "What would make your life not worth living if you were unable to do it?" and "What would you like to be able to do that you cannot do now?" Based on these values, the facilitator helps patients identify their health outcome goals, which are the specific, measurable, actionable, and realistic, and time-bound health and life outcomes (e.g. walk ½ mile daily to visit grandchildren) that patients hope to achieve through their health care, given their care preferences. Care preferences refer to the health care activities (e.g., medications, self-management tasks, health care visits, testing, and procedures) that patients are or are not willing and able to do to achieve their health outcome goals. After the facilitator identifies' the patients' health care priorities, the clinician will work to align clinical decision-making around those priorities during routine clinic visits. This can be manifested by stopping, starting, or continuing therapies in response to knowing the patients' priorities. Patients' priorities will be communicated between care team members via the electronic health record (EHR).

The facilitator and clinicians will be trained in the PPC approach with an initial training, followed by ongoing support from the research team, using quality improvement principles. The investigators will collect the following practice-level data for both PPC-NC and UC clinicians: number of patients, number of encounters, number and type of clinicians, payer mix, and patient demographics of the practices (age, sex, race/ethnicity). The investigators will also collect: socio-demographic factors (age, sex, race/ethnicity, educational level, living arrangement, and marital status), subjective social status, health literacy, and cognitive impairment. A research assistant will collect all patient-reported survey data using the web-based application REDCap (Research Electronic Data Capture) three times over a one year period (baseline, 6 months later, and 12 months post baseline. The investigators will use mixed effects models to compare the primary and secondary patient-reported outcomes between PPC-NC and UC clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 or older
2. Multiple chronic conditions (presence of greater than 2 active health problems) AND either prescribed more than 10 medications or visits to more than two specialists (excluding gynecologists and ophthalmologists) over the past year or have had at least one hospitalization over the past two years
3. Medicare or Medicare-Medicaid eligibility
4. English speaking
5. Current patient with a participating clinician

Exclusion criteria:

1. In hospice or clinician endorsement of a validated palliative care screening question* or clinician responding no to the question that s/he "would not be surprised if the patient passed away within the next 12 months"?
2. End stage renal disease on dialysis
3. Nursing home residence
4. Inability to independently provide informed consent due to dementia or severe psychiatric illness (based on ICD-10 codes or clinician input)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Treatment Burden Score (Baseline to Month 6) | Baseline, Month 6
  Treatment burden will be assessed using the Treatment burden questionnaire- a 15-item measure that assesses the workload imposed by healthcare on patients. Workload includes medication taking, self-monitoring, visits to the provider, laboratory tests, lifestyle changes, and administrative tasks to access and coordinate care. Scoring range is from 0 to 150. Investigators will assess between group change in means of difference in treatment burden score from baseline to month 6. Lower score indicates a worse outcome.
Change in Mean Treatment Burden Score (Baseline to Month 12) | Baseline, Month 12
  Treatment burden will be assessed using the Treatment burden questionnaire- a 15-item measure that assesses the workload imposed by healthcare on patients. Workload includes medication taking, self-monitoring, visits to the provider, laboratory tests, lifestyle changes, and administrative tasks to access and coordinate care. Scoring range is from 0 to 150. Investigators will assess between group change in means of difference in treatment burden score from month 0 to month 12. Lower score indicates a worse outcome.

SECONDARY OUTCOMES:
Change in Mean Shared Decision Making Score (Baseline to Month 6) | Baseline, Month 6
  Investigators will assess shared decision making using the CollaboRATE measure. This 3-item measure assesses the process in which providers and patients work together to make decisions and select treatment. Participants rate, on a scale from 0-9, how much effort was placed into listening, understanding, and including the patient in health care decisions. Lower score indicates a worse outcome.
Change in Mean Shared Decision Making Score (Baseline to Month 12) | Baseline, Month 12
  Investigators will assess shared decision making using the CollaboRATE measure. This 3-item measure assesses the process in which providers and patients work together to make decisions and select treatment. Participants rate, on a scale from 0-9, how much effort was placed into listening, understanding, and including the patient in health care decisions. Investigators will assess between group difference in means of differences in shared decision-making score between baseline and month 6. Lower score indicates a worse outcome.
Change in Electronic Health Record Documentation of Decision-making Based on Patients' Health Priorities (Baseline to Month 12) | Baseline, Month 12
  Investigators will review clinician's notes in the electronic medical record over 12 months of follow-up for documentation of decision-making based on patients' health priorities.
Change in Number of Prescribed Medications (Baseline to Month 6) | Baseline, Month 6
  Investigators will review clinician's notes in the electronic medical record over 12 months of follow-up for documentation of number (percentage) of patients with medications added or stopped over a 12 month period. Investigators will use a data dictionary to guide uniform abstraction.
Change in Number of Prescribed Medications (Baseline to Month 12) | Baseline, Month 12
  Investigators will review clinician's notes in the electronic medical record over 12 months of follow-up for documentation of number (percentage) of patients with medications added or stopped over a 12 month period. Investigators will use a data dictionary to guide uniform abstraction.
Change in Number of Self-Management Tasks | Baseline, Month 12
  Investigators will review clinician's notes in the electronic medical record over 12 months of follow-up for documentation of number (percentage) of patients with self-management tasks added or stopped over a 12 month period. Investigators will use a data dictionary to guide uniform abstraction.
Percentage of Diagnostic Tests, Referrals, and Procedures Ordered or Avoided | Baseline, Month 12
  Investigators will review clinicians' notes in the electronic medical record over 12 months of follow-up for documentation of number (percentage) of patients with diagnostic tests, referrals, or procedures ordered or avoided (defined as mentioned in the electronic health record that they were decided against because they were deemed by the clinician not to be beneficial or unwanted by the patient) over a 12-month period. These measures will be reported in aggregate.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Cené, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - UNC Primary Care of Cary, Cary, North Carolina
  - UNC Family Medicine at Panther Creek, Cary, North Carolina
  - UNC Internal Medicine at Panther Creek, Cary, North Carolina
  - UNC Internal Medicine at Goldsboro, Goldsboro, North Carolina
  - UNC Primary Care at Kenly, Kenly, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: Either IRB, REB or IEC approval and an executed DUA with UNC.

REFERENCES:
- [Result] Tinetti ME, Naik AD, Dindo L, Costello DM, Esterson J, Geda M, Rosen J, Hernandez-Bigos K, Smith CD, Ouellet GM, Kang G, Lee Y, Blaum C. Association of Patient Priorities-Aligned Decision-Making With Patient Outcomes and Ambulatory Health Care Burden Among Older Adults With Multiple Chronic Conditions: A Nonrandomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1688-1697. doi: 10.1001/jamainternmed.2019.4235. PMID 31589281
- See also: Website for Patient Priorities Care — http://patientprioritiescare.org